CLINICAL TRIAL: NCT00604669
Title: Total Parenteral Nutrition(TPN)-Induced Hyperglycemia: Impact on Clinical Outcome in Intensive Care Unit (ICU) and Non-ICU Patients
Brief Title: TPN-Induced Hyperglycemia: Impact on Clinical Outcome in Intensive Care Unit (ICU) and Non-ICU Patients
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Principal Investigator, Emory University
Other Study IDs: IRB00004573; e4573 (Other: Assigned Emory IRB number)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2010-04-07 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-11

CONDITIONS: Hyperglycemia
Keywords: Diabetes; Nutrition/Dietics; clinical outcomes; total parenteral nutrition
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Hyperphagia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A growing body of evidence suggests hyperglycemia is associated with adverse outcomes in patients with and without diabetes. Observational studies document an association between hyperglycemia and poor clinical outcomes in cardiothoracic surgery, elective surgery, myocardial infarction, stroke. Randomized studies indicate glycemic control is associated with improved outcomes in diabetic patients with critically illness. Hyperglycemia is a recognized and common complication of patients receiving total parenteral nutrition (TPN). Few studies in the literature have looked into the impact of TPN-associated inhospital complications and mortality. Accordingly, this study aims to evaluate the impact of hyperglycemia on clinical outcome (infections, systemic sepsis, cardiac complications, acute renal failure, length of stay, and mortality) in patients receiving TPN. We will perform a retrospective chart review of all patients treated with TPN from 1/01/06 to 12/31/06 at Grady Memorial Hospital. We hypothesize that patients receiving TPN who develop hyperglycemia experience higher morbidity (infections, systemic sepsis, cardiac complications, acute renal failure, length of stay) and mortality compared to TPN patients with euglycemia. The results of this study will help us to formulate a prospective randomized clinical trial on the management of TPN-associated hyperglycemia in hospitalized patients.

This study aims to evaluate the impact of hyperglycemia on clinical outcome (infections, systemic sepsis, cardiac complications, acute renal failure, length of stay, in hospital mortality) in patients receiving total parenteral nutrition. We will perform a retrospective chart review of all patients admitted to the hospital receiving TPN from 1/01/06 to 12/31/06 at Grady Memorial Hospital. The results of this study will help us to formulate a prospective randomized clinical trial on the management of TPN-associated hyperglycemia in hospitalized patients.

DETAILED DESCRIPTION:
Hypotheses:

We hypothesize that patients receiving TPN who develop hyperglycemia experience higher morbidity (infections, systemic sepsis, cardiac complications, acute renal failure, length of stay) and mortality compared to TPN patients with euglycemia.

Specific Aim:

To determine the impact of hyperglycemia on clinical outcome (infection, systemic sepsis, cardiac complications, acute renal failure, length of stay, mortality) in patients receiving total parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria: Perform a retrospective chart analysis of all patients receiving TPN at Grady Memorial Hospital during the period of 1/01/06 to 12/31/06.

Exclusion criteria: None except for charts without adequate data sufficient for chart review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving TPN at Grady Memorial Hospital during the period of 1/01/06 to 12/31/06.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University SOM
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 170 charts reviewed
Pre-assignment Details: Nothing to disclose.
Period: Overall Study
Arm/Group | Those Exposed to TPN
Started | 170
Completed | 163
Not Completed | 7
Not completed — lack of information in chart | 7

BASELINE CHARACTERISTICS:
Arm/Group | Those Exposed to TPN
Number analyzed (Participants) | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 120
  >=65 years | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 106
Region of Enrollment [Number; unit: participants]
  United States | 163

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Mortality rate of those with hyperglycemia while on TPN duing the period of 1/01/06 to 12/31/06.
Time Frame: at the end of the chart review of all patients
Measure: Number; unit: mortality rate
Arm/Group | Those Exposed to TPN
Number analyzed (Participants) | 163
mortality rate | 36

ADVERSE EVENTS:
Arm/Group | Those Exposed to TPN
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No